CLINICAL TRIAL: NCT07173192
Title: The Effect of an Individual Empowerment Program Applied to Primary Caregivers of Patients Diagnosed With Schizophrenia on the Burden of Care, Psychological Well-being, and Self-efficacy: A Randomized Controlled Experimental Study
Brief Title: The Effect of an Individual Empowerment Program Provided to Relatives of Schizophrenia Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Zeynep Dag, Servis Hemşiresi, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ARELU-SBF-ZD-01
Record Dates: First submitted 2025-09-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
Keywords: Self Efficacy; Burden, Caregiver; Psychological Well Being; schizophrenia
MeSH Terms: conditions — Schizophrenia; Caregiver Burden; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Data will be collected face-to-face from primary caregivers of patients diagnosed with schizophrenia who are receiving treatment at Istanbul Bakırköy Prof. Dr. Mazhar Osman Mental Health and Neurological Diseases Training and Research Hospital using data collection forms. Individuals who agree to participate in the study and meet the inclusion criteria will be randomized into experimental and control groups. Which caregivers included in the study will be in the intervention group and which will be in the control group will be determined according to the randomization table generated online at https://www.randomizer.org/. Group 1 will be designated as the Intervention Group, and Group 2 will be designated as the Control Group. Data collection tools will be administered to individuals in the experimental and control groups as a pre-test. Individuals in the experimental group will undergo an individual empowerment program consisting of a total of 6 individual empowerment training sessions
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Data collection tools will be administered as a pre-test to individuals in the experimental and control groups. Individuals in the experimental group will receive individual empowerment training sessions as part of a six-session individual empowerment program.
  Interventions: Behavioral: Individual empowerment program
- control group (No Intervention): No intervention will be performed on individuals in the control group; these individuals will receive standard discharge education.

INTERVENTIONS:
Behavioral: Individual empowerment program — Data collection tools will be applied to individuals in the experimental and control groups as a pre-test.
  Individual empowerment training sessions will be applied to individuals in the experimental group totaling (6 sessions) as part of the individual empowerment program. No intervention will be performed on individuals in the control group; they will receive standard discharge education. Data collection tools will be applied to individuals in both groups for post-tests immediately after the experimental group completes all individual empowerment program sessions.
  Arms: experimental group

SUMMARY:
Psychoeducation provided to family members caring for individuals with schizophrenia. Has been found to positively impact caregivers' psychological well-being and the effective management of schizophrenia patients.However, further experimental studies are recommended in this area, along with support for caregivers' psychological well-being. Primary caregivers, which includes both psychoeducation and applications aimed at developing coping skills, on the care burden, psychological well-being,and self-efficacy. Considering the gaps in the literature, the aim of this study is to evaluate the effect of an individual empowerment program applied to primary caregivers of patients diagnosed with schizophrenia on the burden of care, psychological well-being, and self-efficacy.

DETAILED DESCRIPTION:
Schizophrenia is a chronic mental disorder characterized by psychotic experiences accompanied by language, thought, perception, and behavioral disorders, involving periods of relapse and remission (Zhou et al. 2021; Köroğlu et al., 2017). Another definition describes it as a mental illness seen across all segments of society, persisting throughout life with relapses, and leading to impairment in social behavior, personal functioning, and occupational areas (Budiarto et al., 2023; Kırcalı Yılmaz, 2019). Schizophrenia typically begins in late adolescence and early adulthood (Stanley et al. 2017). According to information published on the World Health Organization (WHO) official website in 2022, schizophrenia affects 24 million individuals worldwide, or one in every 300 people (WHO, 2022). This disorder ranks among the top 10 diseases that cause long-term and permanent damage. Its prevalence among individuals aged 15-35 was found to be 0.7% (Çataloluk et al., 2023). The incidence of schizophrenia cases and the recurrence rates of the disease are increasing every year. The World Health Organization (WHO) has shown that recurrence data from 2018 to 2020 has increased from 28% to 54% (Hendro et al., 2024)According to the World Health Organization's (WHO) Mental Health Action Plan 2013-2020, schizophrenia patients generally transition from psychiatric institutions to community-based care once their condition stabilizes (WHO, 2013). As a result of this plan, the development of community-based care for schizophrenia patients, the reduction of mental health hospital capacity without sufficient infrastructure in the community, and the preference for short-term hospital admissions have led to the shift of primary care for schizophrenia patients from the formal health system to families (Chen, 2019; Kırcalı, 2019). Kim et al. (2023) stated in their systematic review and meta-analysis study that approximately 90% of individuals diagnosed with schizophrenia live with family members after being discharged from the hospital. The variable nature of schizophrenia and its debilitating effects create a significant caregiving burden on family caregivers due to the physical, social, emotional, and financial consequences of the illness (Kim et al., 2023, Chen, 2019). Seventy-one point two percent of caregiving families provide an average of 5 hours of care per day (Budiarto et al., 2023). During this process, families also take on additional responsibilities such as managing positive and negative psychiatric symptoms and ensuring adherence to medication treatmentHendro et al., 2024; Zhou et al., 2021; Stanley et al., 2017). As a result of these responsibilities, caregivers may experience difficulties in managing the demands of caregiving. As a result, as seen in numerous studies, caregivers experience high levels of burden (Zhou et al., 2021; Tamizi et al., 2020; Souza et al., 2017), stress, anxiety, depression, neurotic disorders (Tamizi et al., 2020), chronic sadness, stigmatization, and social isolation (Tamizi et al., 2020; Zhou et al., 2021; Souza et al., 2017; Chen et al., 2019)Psychological well-being is a multifaceted concept encompassing individuals' mental health and life satisfaction. This concept includes how individuals feel about themselves, how they find meaning in their lives, and the quality of their social relationships (Çakmakçı, 2023). Psychological well-being is explained by different dimensions such as self-acceptance, establishing positive relationships, autonomy, environmental management skills, life purpose, and personal development (Anastasia & Hardiyanto, 2022; Distina & Kumail, 2019). Family members caring for individuals diagnosed with schizophrenia remain silent about behavioral disorders that involve violence and abuse due to the nature of schizophrenia. Family members neglect their physical and emotional needs while coping with the burden of caregiving (Nuraini et al., 2023; Ehsan et al., 2018). This negatively affects the psychological well-being of caregivers (Hendro et al., 2024; Nuraini et al., 2023; Sharma et al., 2021). Research in the literature has shown that psychological well-being decreases as the caregiving burden increases (Thongthammarat et al., 2022; Sharma et al., 2021). In their study investigating the negative effects of caregiving burden, Ehsan et al. (2018) reported that caregivers of schizophrenia patients had psychological well-being that was 2 times lower and a depression risk that was 7 times higher compared to healthy individualsThese findings reveal that caregivers are at risk for mental illness and require special support from other family members, the community, and healthcare providers.

These findings reveal that caregivers are at risk for mental illness and require special support from other family members, the community, and healthcare providers. Zimmerman (1981) defined self-efficacy as "an individual's judgments about their ability to accomplish and succeed in a task." Self-efficacy is an individual's beliefs and judgments about their capacity to overcome difficult situations they may encounter in the future (Fitzgeraldson et al., 2024; Durmaz, 2011). Another definition describes it as the belief in oneself during the process of achieving a desired outcome (Ebrahem et al., 2024). An increase in an individual's perception of self-efficacy leads to the display of positive health behaviors.Low self-efficacy feelings can lead to low self-esteem and pessimism in individuals, while high self-efficacy feelings encourage overcoming difficulties and working towards goals (Durmaz et al., 2014).

The caregiver's internal motivation is one of the determining factors affecting the burden of care.

Being able to manage the symptoms of schizophrenia during the care process and cope with difficulties is of great importance for both patients and caregivers.

Ebrahem et al. (2024) examined the relationship between self-efficacy, care burden, and hope among caregivers of individuals with psychotic disorders. In a study by Ebrahem et al. (2024) examining the relationship between self-efficacy, care burden, and hope among caregivers of individuals with psychotic disorders, the self-efficacy levels of individuals caring for chronic psychotic illnesses were found to be low to moderate.

Reviewing the literature, other studies have found a negative correlation between care burden and self-efficacy.

That is, as care burden increases, caregivers' self-efficacy levels are found to be low (Ebrahem et al., 2024; Ramzani et al., 2019; Durmaz et al., 2014; Durmaz, 2011).Thongthammarat et al. (2022) examined the effectiveness of an enhanced psychological well-being intervention on the psychological well-being and care burden of family members caring for individuals with schizophrenia. Their study found that an enhanced psychological well-being intervention provided to relatives of individuals diagnosed with schizophrenia increased the psychological well-being levels of these relatives and also reduced their care burden.

Ebrahem et al. (2024) examined the relationship between self-efficacy, care burden, and hope among caregivers of individuals with psychotic disorders. Their study found that as the care burden increased among caregivers of individuals with psychotic disorders, their levels of self-efficacy decreased.The individual empowerment program includes a series of activities and strategies aimed at helping individuals discover their potential, develop their talents, and improve their quality of life. These types of programs are designed to empower individuals psychologically, socially, and economically. In particular, individual empowerment increases individuals' ability to make their own decisions, strengthens their self-confidence, and develops their ability to cope with difficulties in their lives (Krenz et al., 2013; Setyoadi et al., 2023). These programs aim to reduce the stress and difficulties experienced by patients' relatives, improve their psychosocial health, and increase their overall quality of life. (Ercan et al., 2019; Harmancı, 2016). In this context, the educational and counseling roles of psychiatric nurses toward families are critically important in reducing the burden on caregivers and developing coping mechanisms (Kaya, 2018; Gök et al., 2023). Individual empowerment programs implemented by psychiatric nurses are an important support mechanism for relatives of schizophrenia patients. These programs improve the knowledge and skills of relatives, develop their ability to cope with stress, and improve their overall quality of life (Dost, 2023; Buldukoğlu et al., 2011).It is recommended that psychiatric nurses provide education and counseling that includes coping strategies to help caregivers of individuals with psychotic disorders improve their self-efficacy (Ebrahem et al., 2024). Additionally, it has been noted that more interventional research is needed, including specialized interventions that incorporate skill development and psychoeducation for the care of schizophrenia patients, to alleviate the care burden on family members caring for schizophrenia patients (Thongthammarat et al., 2022). Psychoeducation provided to family members caring for individuals with schizophrenia has been found to have positive effects on caregivers' psychological well-being and the effective management of individuals with schizophrenia; however, more experimental studies on this topic and support for caregivers' psychological well-being are recommended (Sharma et al., 2021; Ehsan et al., 2018). Furthermore, since the studies in the literature were group studies, Kim et al. (2023) recommended that future interventions be applied individually in their meta-analysis examining the effectiveness of interventions for relatives of schizophrenia patients.No interventional studies have been found examining the effects of an individual empowerment program for patients diagnosed with schizophrenia that includes both psychoeducation and coping skills training for primary caregivers on the burden of care, psychological well-being, and self-efficacy. Considering the gaps in the literature, the aim of this study is to evaluate the effect of an individual empowerment program applied to primary caregivers of patients diagnosed with schizophrenia on the burden of care, psychological well-being, and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

Being the primary caregiver of a patient diagnosed with schizophrenia and other psychotic disorders Volunteering to participate in the study Being 18 years of age or older Being literate Not having a psychiatric illness (diagnosis) Not having a serious mental or physical disorder that prevents communication

Exclusion Criteria:

Providing care to patients with severe organic brain syndrome such as alcohol or substance dependence, intellectual disability, dementia, or delirium, or with a previous or current general medical condition that could impair cognitive function Withdrawal from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
The psychological well-being scale based on the individual empowerment program will be used to measure the care burden of individuals providing primary care to those diagnosed with schizophrenia. (time frame: 6 week) | 6 week
  The training will be conducted in person.
The care burden scale based on the individual empowerment program will be used to measure the care burden for individuals providing primary care to individuals diagnosed with schizophrenia. (Time frame: 6 weeks) | 6 week
  Face-to-face training will be provided.
The self-efficacy scale based on the individual empowerment program will be used to measure the care burden of individuals providing primary care to people diagnosed with schizophrenia. (time frame: 6 weeks) | 6 week
  The training will be conducted in person.

CONTACTS AND LOCATIONS:
Overall Officials: zeynep dağ psychiatric nurse, Principal Investigator — Istanbul Arel University
Locations (1):
- Istanbul Arel University, Istanbul, Cevizlibağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I'm not sure